CLINICAL TRIAL: NCT03516214
Title: An Open-label, Multicenter, Phase I Dose-escalation Trial of EGF816 and Trametinib in Patients With Non-small Cell Lung Cancer and Acquired EGFR p.T790M-positive Resistance to 1st or 2nd Generation EGFR TKI Therapy Remark: According to Version V02_0 of the Protocol, Patients May Also be Eligible if EGFR TKI-treatment naïve, EGFR p.T790M-negative at Progression While on EGFR TKI Therapy or After Progression While on Osimertinib Treatment
Brief Title: EGF816 and Trametinib in Patients With Non-small Cell Lung Cancer Harboring Activating EGFR Mutations
Acronym: EATON
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Juergen Wolf, Prof. Dr., University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1784; 2016-003944-35 (EudraCT Number); AIO-TRK-0216 (Other: Arbeitsgemeinschaft Internistische Onkologie)
Record Dates: First submitted 2018-03-29; First posted 2018-05-04 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Bronchial Neoplasms
Keywords: acquired resistance; EGFR p.T790M-positive; osimertinib resistance; EGFR p.T790M-negative
MeSH Terms: conditions — Bronchial Neoplasms | interventions — nazartinib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EGF816 (nazartinib) and trametinib (Experimental): Patients will receive oral EGF816 (nazartinib) and trametinib at escalating dose levels. Intra-patient dose-escalation will not be allowed.
  Interventions: Drug: EGF816; Drug: Trametinib

INTERVENTIONS:
Drug: EGF816 — Continuous oral treatment (once daily) with the 3rd generation EGFR inhibitor EGF816.
  Other Names: Nazartinib
Drug: Trametinib — Continuous oral treatment (once daily) with the MEK inhibitor trametinib.
  Other Names: Mekinist

SUMMARY:
The aim of this trial is to identify the maximum tolerated dose (MTD)/recommended phase II dose (RP2D), to define pharmacokinetic (PK) parameters and the preliminary efficacy of a continuous treatment with EGF816 and trametinib in locally advanced or metastatic (stage IIIB or IV) lung cancer patients with activating mutations in the epithelial growth factor receptor (EGFR).

DETAILED DESCRIPTION:
The population of interest for this trial is defined by patients with non-small cell lung cancer (NSCLC) harbouring the sensitizing EGFR mutations del19 or p.L858R. Patients may be enrolled in first- or later lines of therapy and independently of the prior (approved) EGFR inhibitor administered and independently of the EGFR p.T790M-status. Those individuals whose tumors harbour high-level amplifications of MET or other EGFR mutations except for del19, p.L858R or p.T790M will be excluded from the trial. The molecular status must have been determined in a biopsy collected at progression to the last systemic and prior to the initiation of the trial treatment

The aim of the trial is to identify the maximum tolerated dose (MTD)/recommended phase II dose (RP2D) for a continuous treatment with the 3rd generation EGFR inhibitor EGF816 and the MEK inhibitor trametinib.

The recommendations for dose level escalations will be based on an "up-and-down" design proposed by Storer, 1989. The dose limiting toxicity (DLT) period comprises the first 28 days of treatment with EGF816 and trametinib at the designated dose level (Cycle 1).

PK parameters of the combination treatment will be assessed for every dose level in every patient during the dose-escalation part.

Preliminary efficacy of EGF816 and trametinib in the trial population will be assessed by RECIST (v1.1) analysis of scheduled CT scans (every 8 weeks or as clinically indicated.

Throughout the study blood samples will be collected to monitor cell free plasma DNA (cfDNA).

Patients who develop resistance upon treatment with the study drugs will undergo a rebiopsy to identify potential mechanisms of resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must have been obtained prior to any screening procedures.
2. Patients (male or female) ≥ 18 years of age.
3. Histologically documented, locally advanced or recurrent (stage IIIB who are not eligible for combined modality treatment) or metastatic (stage IV) non-small cell lung cancer.
4. Presence of at least one measurable lesion according to RECIST v.1.1.
5. ECOG performance status ≤ 2
6. Patients must have NSCLC harbouring EGFR p.L858R or EGFR del19 as assessed by local testing.
7. Patients must be EGFR TKI treatment naïve (prior chemotherapy treatment is allowed) or must have progressed while on continuous treatment with a first- or second-generation EGFR TKI (EGFR p.T790M-negative or -positive) or must have progressed while on continuous treatment with osimertinib (EGFR p.T790M-negative or -positive)
8. In patients who have received no prior EGFR TKI treatment, an archival biopsy sample, defined as a sample being obtained prior to any anti-cancer treatment is mandatory. If an archival biopsy fulfilling this criterion is not available, patients must be suitable and willing to undergo baseline biopsy according to the local institution's guidelines (newly obtained biopsy).
9. In patients who have received prior EGFR TKI treatment, an archival biopsy sample, defined as a sample being obtained after or during progression upon the last anti-cancer treatment is mandatory. No consecutive line of treatment must have been given after collection of the rebiopsy and inclusion into this trial. If an archival rebiopsy fulfilling these criteria is not available, patients must be suitable and willing to undergo baseline biopsy according to the local institution's guidelines (newly obtained biopsy).
10. In patients who have received prior EGFR TKI treatment, EGFRp.T790M mutation status must have been assessed by local testing in the tumour sample fulfilling the requirements of inclusion criterion 9.
11. Patients who have received prior osimertinib treatment, may only be eligible if no standard treatment approach outside this trial is available or feasible (e.g. chemotherapy)
12. Patients who have progressed while on continuous treatment with a first- or second-generation EGFR inhibitor and whose tumour has been tested EGFR p.T790M-negative may only be eligible if no standard treatment approach outside this trial is available or feasible (e.g. chemotherapy).
13. In patients who have received prior EGFR TKI treatment, progression of disease according to RECIST v1.1 while on continuous treatment with an EGFR TKI (e.g. erlotinib, gefitinib, afatinib or osimertinib) must be documented.

Exclusion Criteria:

1. History of allergic reactions or hypersensitivity to one of the study drugs or to any component of the study drugs
2. Prior treatment with any investigational agent known to inhibit EGFR (mutant or wild-type)
3. Prior treatment with any agent known to inhibit MEK/ERK or other mediators of RAS pathway.
4. Patients with high level MET amplification in the archival or newly obtained biopsy sample as determined by local testing. High-level MET amplification is defined as: a) a MET/CEN7 ratio ≥2.0 and/or b) an average MET gene copy number per cell of ≥6.0 [modified Schildhaus et al., 2015].
5. Patients with EGFR mutations other than EGFR del19, p.L858R or p.T790M.
6. Patients with brain metastases. However, if radiation therapy and/or surgery has been completed at least 4 weeks prior to screening for the trial and evaluation by CT (with contrast enhancement) or MRI at study baseline demonstrates the disease to be stable and if the patient remains asymptomatic and off steroids, then patients with brain metastases may be enrolled.
7. Patients with presence or history of carcinomatous meningitis.
8. Any acute or chronic medical, mental or psychological condition, which in the opinion of the investigator would not permit the patient to participate or complete the study or understand the patient information
9. History of hepatitis B (HBV) or hepatitis C (HCV) or positive result in mandatory testing for acute or chronic hepatitis B or hepatitis C
10. Known HIV infection or history of HIV infection independent from the cellular immune status
11. Patients who receive any continuous, long term immunosuppressive treatment, including long term treatment with steroids at immunosuppressive doses at the time of study entry
12. Patients who underwent bone marrow or solid organ transplantation, including patients who do not receive any immunosuppressive treatment.
13. Presence or history of any other primary malignancy other than NSCLC within 5 years prior to enrolment into the trial. Except from this: Adequately treated basal or squamous cell carcinoma of the skin or any adequately treated in situ carcinoma
14. Any of the following within 6 months prior to first trial drug administration: Myocardial infarction (NSTEMI or STEMI), severe/unstable angina pectoris, symptomatic congestive heart failure (> NYHA II), uncontrolled hypertension, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack, atrial fibrillation of CTCAE Grade ≥ 2, ongoing cardiac dysrhythmias of CTCAE Grade ≥ 2, including corrected QTcF prolongation of > 480 ms,
15. Aortic valve stenosis with mean gradient ≥ 25 mmHg and aortic valve area of ≤ 1.5 cm2
16. Any other cardiac valve abnormality of more than mild degree/stage
17. Left ventricular ejection fraction (LVEF) of < 50 %
18. History of congenital long QT-syndrome or Torsades de Pointes
19. History of retinal vein occlusion (RVO) or retinal pigment epithelial detachment (RPED)
20. Unable or unwilling to swallow tablets or capsules
21. Patients with impaired gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of EGF816 (e.g., ulcerative diseases, uncontrolled nausea, vomiting diarrhoea, or malabsorption syndromes
22. Patients have received anticancer treatment within the following time frames prior to the first dose of study treatment:

    1. Conventional cytotoxic chemotherapy: ≤ 4 weeks (≤ 6 weeks for nitrosoureas, mitomycin-C and suramin)
    2. Biological therapy (e.g., antibodies, excluding PD-1 or PD-L1 antibodies): ≤ 4 weeks
    3. PD-1/PD-L1 antibodies (e.g., nivolumab, pembrolizumab): ≤ 5 half-times
    4. Non-cytotoxic anti-cancer therapeutic (e.g., tyrosine kinase inhibitors): ≤ 5 half-times or ≤ 1 weeks (whichever is longer)
    5. Other investigational agent: ≤ 4 weeks
    6. Radiation therapy (excluding palliative radiation, e.g., of bone metastases): ≤ 4 weeks
    7. Major surgery (excluding minor surgical interventions, e.g., vascular device implantation): ≤ 2 weeks
23. Laboratory values as listed below, that cannot be corrected to normal limits within screening :

    1. Absolute Neutrophil Count (ANC) < 1.5 x 10^9/L
    2. Haemoglobin (Hb) < 9 g/dL
    3. Platelets (PLT) < 100 x 10^9/L
    4. Total bilirubin > 1.5 x upper limit of normal (ULN). For patients with confirmed Gilbert's disease total bilirubin > 2.5 x ULN
    5. AST and/or ALT > 3 x ULN
    6. AST and/or ALT > 5 x ULN in patients with liver involvement
    7. Serum creatinine > 1.5 x ULN
    8. Measured or calculated creatinine clearance ≤ 45 mL/min
    9. Serum amylase and/or lipase CTCAE Grade > 2
    10. Potassium, magnesium, phosphorus, total calcium (corrected from serum albumin) > ULN
24. Patients receiving treatment with any medication that are known to be

    1. Strong inhibitors or inducers of CYP3A4/5
    2. Substrates of CYP2D6 with narrow therapeutic index
    3. and that cannot be discontinued at least 7 days prior to the first dose of the study drugs.
    4. For further information please refer to Section 11.7 and the Concomitant Medication Manual.
25. Patients with a history of or presence of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis
26. Pregnancy or breastfeeding/nursing women
27. Women of child-bearing potential (for definition see Section 8.3.3) unless they use highly effective methods of contraception during treatment and for four months after withdrawal of study treatment (for methods of contraception see Section 8.3.4)
28. Sexually active males unless they use a condom during intercourse for the time of study treatment and for four months after the withdrawal of study treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting-toxicities (DLT) of the combination of EGF816 and trametinib to assess the maximum tolerated dose (MTD)/recommended phase II dose (RP2D) | Approximately one and a half years (from FPFV until the end of the DLT period of the last patient included into the trial or until death of the last patient, whichever occurs first)
  Incidence of dose-limiting-toxicities (DLT) that occur during the DLT period (i.e. first 4 weeks of treatment) of each patient in the dose-escalation part (N=18)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | Approximately four years (from FPFV until the completion of the clinical trial)
Number of patients who experienced dose interruptions or reductions | Approximately four years (from FPFV until the end-of-treatment visit of the last patient or until death of the last patient, whichever occurs first)
Objective response rate (ORR) according to RECIST 1.1 | Approximately 4 years (from FPFV until the progression of the last patient treated within the trial or until death of the last patient, whichever occurs first)
Disease control rate (DCR) according to RECIST 1.1 | Approximately 4 years (from FPFV until the progression of the last patient treated within the trial or until death of the last patient, whichever occurs first)
Progression-free survival (PFS) according to RECIST 1.1 | Approximately 4 years (from FPFV until the progression of the last patient treated within the trial or until death of the last patient, whichever occurs first)
Duration of response (DOR) according to RECIST 1.1 | Approximately 4 years (from FPFV until the progression of the last patient treated within the trial or until death of the last patient, whichever occurs first)
Time to response (TTR) according to RECIST 1.1 | Approximately 4 years (from FPFV until the progression of the last patient treated within the trial or until death of the last patient, whichever occurs first)
overall survival (OS) | Approximately 4 years (from FPFV until the progression of the last patient treated within the trial or until death of the last patient, whichever occurs first)
Plasma concentration vs time profiles - plasma PK parameters of EGF816 and trametinib | Approximately two years (from FPFV until the completion of four months of treatment of the last patient or until death of the last patient, whichever occurs first)

OTHER OUTCOMES:
Massively parallel sequencing (MPS), FISH and phospho-immunoblots of pre-treatment tumour samples in order to assess potential predictive markers for response and resistance | Approximately one and a half years (from FPFV until the inclusion of the last patient)
Massively parallel sequencing (MPS), FISH and phospho-immunoblots of post-treatment tumour samples in order to assess potential predictive markers for response and resistance | Approximately four years (from the first progressing patient until the last progressing patient or death of the last patient, whichever occurs first)
MPS of cell-free DNA (cfDNA) at baseline, during treatment and at progression to assess the value of cell-free plasma DNA (cfDNA) for assessment of predictive molecular markers of response and resistance and for monitoring patients under therapy | Approximately four years (from FPFV until the progression of the last patient or death of the last patient, whichever occurs first)
Establishment of conditionally reprogrammed tumour cells (CRCs) from fresh tumour tissue for the study of resistance mechanisms and drug sensitivity | Approximately four years (from the first progressing patient until the last progressing patient or death of the last patient, whichever occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Wolf, Prof. Dr., Principal Investigator — University Hospital of Cologne
Locations (7):
- Germany (5):
  - University Hospital of Cologne, Cologne
  - University Hospital Dresden, Dresden
  - University Hospital Essen, Essen
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Würzburg, Würzburg
- Spain (2):
  - Instituto Oncológico Dr. Rosell, Barcelona
  - Vall d'Hebron University Hospital, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided